CLINICAL TRIAL: NCT01544439
Title: The Efficacy of Occlusal Stabilization Appliance Associated to Counseling in the Management of Myofascial Pain Chronic and in the Improvement of the Quality of Life of Patients With Temporomandibular Disorders
Brief Title: Occlusal Splint and Counseling to Temporomandibular Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Patra-cia Rocha Coelho (Other)
Collaborators: Federal University of Juiz de Fora (Other)
Responsible Party: Sponsor-Investigator, Patra-cia Rocha Coelho, Principal Investigator, Federal University of Juiz de Fora
Organization: Federal University of Juiz de Fora (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTN: U111-1128-3875; 0183.0.180.000-11 (Registry Identifier: Comissão Nacional de Ética em Pesquisa (CONEP)); 199/2011 (Registry Identifier: Committee on Ethics in Human Research of Federal University of Juiz de Fora)
Record Dates: First submitted 2012-02-23; First posted 2012-03-06 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-03

CONDITIONS: Temporomandibular Disorders; Stress Psychological; Musculoskeletal Diseases
Keywords: Temporomandibular joint disorders; Stress psychological; Depression; Quality of Life
MeSH Terms: conditions — Temporomandibular Joint Disorders; Stress, Psychological; Musculoskeletal Diseases; Depression | interventions — Splints; Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral stabilization appliance,counselling (Experimental): The reversible occlusal therapy by stabilizing appliance used by patients in Study Group shall be made by the same dental technician and will be adjusted by the same dentist, therapist represented by the researcher. Will be played simultaneous occlusal contacts in centric relation position and malocclusion by canine and protrusive guides. Patients receive oral and written instructions about self-care (counseling), including, in addition to instructions on their condition of TMD and an explanation of the possible factors that contribute to the etiology of the same.
  Interventions: Procedure: stabilizing appliance
- Non-occluding splint, counselling (Placebo Comparator): The non-occlusive splint (placebo) will also be made by the same dental technician. They differ by the plates did not interfere with the occlusal tooth gear, ie, do not alter the position of closing jaws. As not lead acrylic on the occlusal surfaces of teeth, adequate retention is given by an arch wire in orthodontic buccal surface of teeth. All patients will submitted a counseling approach / self-care. Patients receive oral and written instructions about self-care, including, in addition to instructions on their condition of TMD and an explanation of the possible factors that contribute to the etiology of the same.
  Interventions: Procedure: Non-occluding splint, counseling

INTERVENTIONS:
Procedure: stabilizing appliance — The reversible occlusal therapy be made by the same dental technician and will be adjusted by the same dentist, therapist represented by the researcher. Will be played simultaneous occlusal contacts in centric relation position and malocclusion by canine and protrusive guides. The patients will be assessed at weekly intervals (between the query and the following board installation) and then biweekly during the period of 90 days. There shall be a gradual reduction in the daily use of the plate, and the first two weeks the device is indicated for 24 hours a day, being removed only for eating and cleaning. At each visit clinical follow-up, shall be established a gradual reduction in the time of use so that the last three weeks of treatment are achieved 8h/day use.
  Other Names: Occlusal stabilization appliance; Oral splints; Stabilization splint theraphy
  Arms: Oral stabilization appliance,counselling
Procedure: Non-occluding splint, counseling — The non-occlusive splint (placebo) will also be made by the same dental technician. They did not interfere with the occlusal tooth gear, ie, do not alter the position of closing jaws. They are adjusted based on the verification of the occlusion, so that the card does not interfere with movements or maximum intercuspation excursive lateral and protrusion, so that only the patient's teeth come into contact, without interference from the resin and the acrylic staple . The assessment of these patients occur at the same intervals recommended for patients in the experimental group being established on the same treatment protocol with respect to the daily use of the splint.
  Other Names: Splint control; Nonsplint therapy
  Arms: Non-occluding splint, counselling

SUMMARY:
The aim of this study was to evaluate the effectiveness of the splint occlusal associated with counseling in reducing pain in patients with temporomandibular disorders, under the assumption that the occlusal appliance offers the highest rates of improvement than their placebo.

DETAILED DESCRIPTION:
* The aim of this double-blind randomized control trial was to evaluate the efficacy of occlusal stabilization appliance associated to counseling in the management of myofascial pain chronic and in the improvement of the quality of life of patients with temporomandibular disorders (TMD).
* In order to reduce the likelihood of systematic errors and allow the use of statistical tests is used randomization processes or randomization of the volunteers in the different groups from a sequence generated by a specific program (Randomization.com), and the principal investigator masked for this division. For this, a second researcher, appointed to undertake the division of patients into groups that maintain confidential information from groups and their participants, revealing only the researcher therapist at the time of first therapy session. The number of individuals randomized to the experimental group will be equal to the control group.

  1. Study Group Intervention The reversible occlusal therapy by stabilizing appliance used by patients in Study Group shall be made by the same dental technician and will be adjusted by the same dentist, therapist represented by the researcher. Will be played simultaneous occlusal contacts in centric relation position and malocclusion by canine and protrusive guides. The patients will be assessed at weekly intervals (between the query and the following board installation) and then biweekly during the period of 90 days. There shall be a gradual reduction in the daily use of the plate, and the first two weeks the device is indicated for 24 hours a day, being removed only for eating and cleaning. At each visit clinical follow-up, shall be established a gradual reduction in the time of use so that the last three weeks of treatment are achieved 8h/day use.
  2. Control Group Intervention The non-occlusive splint (placebo) will also be made by the same dental technician. They differ by the plates did not interfere with the occlusal tooth gear, i.e., do not alter the position of closing jaws. As not lead acrylic on the occlusal surfaces of teeth, adequate retention is given by an arch wire in orthodontic buccal surface of teeth. They are adjusted based on the verification of the occlusion, so that the card does not interfere with movements or maximum intercuspation excursive lateral and protrusion, so that only the patient's teeth come into contact, without interference from the resin and the acrylic staple . The assessment of these patients occur at the same intervals recommended for patients in the experimental group being established on the same treatment protocol with respect to the daily use of the plate.
* In this study, all patients (study and control group) will undergo a counseling approach/self-care. Patients receive oral and written instructions about self-care, including, in addition to instructions on their condition of TMD and an explanation of the possible factors that contribute to the etiology of the same. The program also includes self-care guidelines on the use of moist heat or ice, use of soft diet, reduction of parafunctional habits (such as clenching and grinding your teeth or chewing gum), holding the rest of the postural position of the jaw (teeth apart , lips and tongue touching slightly pushing the front teeth), performing simultaneous bilateral chewing and modify posture to sleep. This approach will be reinforced verbally at each subsequent session.

ELIGIBILITY:
Inclusion Criteria:

All subjects participated in this study volunteers by signing the consent form. Inclusion criteria are as follows:

* female subjects;
* aged 20 to 55 years;
* irrespective of race, social status or religion;
* presence of pain intensity of at least moderate (at least 4.0 on VAS), shown in the first clinical assessment;
* diagnosis of myofascial pain persisting for a minimum period of six months.

Exclusion Criteria:

* history of psychiatric disorders or treatment for neurological or psychological disorders;
* volunteers with severe intellectual or physical disability that would hinder the collection of data;
* history of systemic diseases that generate joint symptoms, muscle or rheumatologic, such as rheumatoid arthritis and fibromyalgia;
* pain attributed to a well-defined local cause, such as pulpitis, trigeminal neuralgia and cancer pain;
* attributable to migraine pain or infection;
* report of any previous treatment for TMD;
* treatment with drugs affecting the central nervous system (muscle relaxants, anticonvulsants, opioids, and antidepressants) and treatment with analgesics and anti-inflammatory drugs, with or without prescription, concomitant therapies to be instituted in this research;
* report of facial trauma as a possible etiology of TMD;
* subject denture wearers an upper or lower;
* volunteers aged under 20 or over 55 years;
* male individuals.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of physical symptoms | Participants will be monitored during the study period to assess changes in physical symptoms at 12 weeks.
  The measurement of spontaneous orofacial pain intensity will be obtained through the Visual Analogue Scale (VAS). Evaluated before and after three months of interventions, will be obtained from the average intensity of pain experienced by each group. The evolution of physical symptoms reported in each group will verify the effectiveness of interventions instituted in each group.
Assessment of Quality of Life related to TMD | Participants will be monitored during the study period to assess changes in quality of life in 12 weeks
  The comparison of scores in the two periods indicate a possible change in the index of quality of life. The instrument used for this will be the profile of the Oral Health Impact (OHIP-14).

SECONDARY OUTCOMES:
Evaluation of psycho-emotional aspects related to the TMD | The psycho-emotional aspects will be evaluated before and after the intervention period of three months (12 weeks) to initiation of therapy
  The Diagnostic Criteria for Research of temporomandibular disorders (RDC / TMD, Axis II)will be used. To assess the impact of psycho TMD, we investigate measures of depression and nonspecific physical symptoms accompanied by pain (somatization).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia R. Coelho, Master, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- Federal University of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

REFERENCES:
- [Result] Alencar F Jr, Becker A. Evaluation of different occlusal splints and counselling in the management of myofascial pain dysfunction. J Oral Rehabil. 2009 Feb;36(2):79-85. doi: 10.1111/j.1365-2842.2008.01913.x. Epub 2008 Oct 22. PMID 18976268
- [Result] Dao TTT, Lavigne GJ, Charbonneau A, Feine JS, Lund JP. The efficacy of oral splints in the treatment of myofascial pain of the jaw muscles: a controlled clinical trial. Pain. 1994 Jan;56(1):85-94. doi: 10.1016/0304-3959(94)90153-8. PMID 8159444
- [Result] De Laat A, Stappaerts K, Papy S. Counseling and physical therapy as treatment for myofascial pain of the masticatory system. J Orofac Pain. 2003 Winter;17(1):42-9. PMID 12756930
- [Result] Ekberg E, Vallon D, Nilner M. The efficacy of appliance therapy in patients with temporomandibular disorders of mainly myogenous origin. A randomized, controlled, short-term trial. J Orofac Pain. 2003 Spring;17(2):133-9. PMID 12836501
- [Result] Jokstad A, Mo A, Krogstad BS. Clinical comparison between two different splint designs for temporomandibular disorder therapy. Acta Odontol Scand. 2005 Aug;63(4):218-26. doi: 10.1080/00016350510019982. PMID 16040444
- [Result] Riley JL 3rd, Myers CD, Currie TP, Mayoral O, Harris RG, Fisher JA, Gremillion HA, Robinson ME. Self-care behaviors associated with myofascial temporomandibular disorder pain. J Orofac Pain. 2007 Summer;21(3):194-202. PMID 17717958
- [Result] Truelove E, Huggins KH, Mancl L, Dworkin SF. The efficacy of traditional, low-cost and nonsplint therapies for temporomandibular disorder: a randomized controlled trial. J Am Dent Assoc. 2006 Aug;137(8):1099-107; quiz 1169. doi: 10.14219/jada.archive.2006.0348. PMID 16873325
- [Result] Wright E, Anderson G, Schulte J. A randomized clinical trial of intraoral soft splints and palliative treatment for masticatory muscle pain. J Orofac Pain. 1995 Spring;9(2):192-9. PMID 7488989
- See also: Page SISNEP where they found information about the submission and approval of the study to the Platform Brazil - the Ethics in Human Research - Dean of Research / UFJF — http://portal2.saude.gov.br/sisnep/extrato_projeto.cfm?CODIGO=443975